CLINICAL TRIAL: NCT04734730
Title: Phase II Study of Talazoparib With Androgen Deprivation Therapy and Abiraterone in Castration Sensitive Prostate Cancer
Brief Title: Talazoparib With Androgen Deprivation Therapy and Abiraterone for the Treatment of Castration Sensitive Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20476; NCI-2020-10199 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20476 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; bicalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin; Leuprolide; luprolide acetate gel depot; Prednisone; deltacortene; prednylidene; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (talazoparib, androgen deprivation therapy) (Experimental): Patients receive talazoparib PO QD, abiraterone acetate PO QD, and prednisone PO QD on days 1-28. Patients also receive androgen deprivation therapy consisting of degarelix SC on day 1; leuprolide acetate IM on day 1 and bicalutamide PO QD on days 1-28 of cycle 1 and then leuprolide acetate IM on day 1 of subsequent cycles; leuprolide acetate IM on day 1 and bicalutamide PO QD on days 1-28 of cycle 1 and then leuprolide acetate IM on day 1 of cycles 2, 5, 8, and 11; or goserelin acetate SC monthly or every 3 months. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Bicalutamide; Drug: Degarelix; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Drug: Prednisone; Other: Questionnaire Administration; Drug: Talazoparib

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Questionnaire Administration — Ancillary studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase II trial studies the effect of talazoparib with androgen deprivation therapy and abiraterone in treating castration sensitive prostate cancer patients. Talazoparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Androgen can cause the growth of prostate tumor cells. Degarelix, leuprolide acetate, bicalutamide, goserelin acetate, and abiraterone lowers the amount of androgen made by the body. This may help stop the growth of tumor cells that need androgen to grow. Giving talazoparib with androgen deprivation therapy and abiraterone may improve cancer control for patients with castration sensitive prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Increase the efficacy of first-line therapy for men with metastatic castration-sensitive prostate cancer by adding the PARP inhibitor talazoparib to standard therapy with androgen deprivation therapy (ADT) + abiraterone acetate (abiraterone).

II. Study the efficacy of abiraterone and talazoparib in an ethnically diverse population.

III. Evaluate whether androgen receptor genetic variation may identify a subpopulation of patients who benefit, even in the absence of homologous repair deficiency mutations.

OUTLINE:

Patients receive talazoparib orally (PO) once daily (QD), abiraterone acetate PO QD, and prednisone PO QD on days 1-28. Patients also receive androgen deprivation therapy consisting of degarelix subcutaneously (SC) on day 1; leuprolide acetate intramuscularly (IM) on day 1 and bicalutamide PO QD on days 1-28 of cycle 1 and then leuprolide acetate IM on day 1 of subsequent cycles; leuprolide acetate IM on day 1 and bicalutamide PO QD on days 1-28 of cycle 1 and then leuprolide acetate IM on day 1 of cycles 2, 5, 8, and 11; or goserelin acetate SC monthly or every 3 months. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologically or cytologically proven diagnosis of adenocarcinoma of the prostate. (Note: Gleason score not required if biopsy of metastasis was used to make the histologic diagnosis)
* All patients must have metastatic disease: either soft tissue and/or bony metastases prior to initiation of androgen. Measurable disease is not required
* Baseline imaging must have been performed within 42 days before or 14 days after initiating luteinizing hormone releasing hormones (LHRH) therapy. All disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients may have started on LHRH therapy for metastatic prostate cancer provided this was initiated no longer than 60 days prior to registration

  * Patients may have received neoadjuvant and/or adjuvant LHRH therapy during definitive treatment or salvage radiation; if so at least 12 months must have elapsed from the last LHRH injection and baseline testosterone must be > 150 ng/dL
  * No restriction on bicalutamide used for flare prevention or combined therapy however bicalutamide must be stopped at registration
* Patients must have a Karnofsky performance status of 60 - 100
* Men of reproductive potential and those who are surgically sterilized (i.e., vasectomy) must agree to practice effective barrier contraception or agree to abstain from intercourse while receiving treatment on this study and for at least 4 months after protocol treatment ends
* Bilirubin =< 2 x institutional upper limit of normal (ULN) (obtained within 28 days prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x institutional ULN, or =< 5 x institutional ULN if liver metastases are present (obtained within 28 days prior to registration)
* Calculated creatinine clearance >= 30 mL/min using a serum creatinine obtained within 28 days prior to registration
* Leukocytes >= 3,000/mcL (obtained within 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained within 28 days prior to registration)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to registration)
* Platelets >= 100,000/mcL (obtained within 28 days prior to registration)
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients may have received prior androgen deprivation therapy (ADT) -neoadjuvant and/or adjuvant, or in conjunction with salvage radiation - but it must not have lasted for more than 36 months. Single or combination therapy allowed. At least 6 months must have elapsed since completion of androgen deprivation therapy in the neoadjuvant and/or adjuvant setting, and serum testosterone must be > 150 ng/mL within 28 days prior to registration. Note: Serum testosterone assessment is required for eligibility for only those with prior treatment with ADT

  * Patients who have already started on LHRH therapy are eligible, provided no more than 60 days have elapsed from LHRH injection (or surgical castration) for metastatic prostate cancer prior to registration. The start date of medical castration is considered the day the patient first received an injection of a LHRH agonist/antagonist (or orchiectomy), not an oral antiandrogen. Subjects may not already be taking abiraterone, enzalutamide, apalutamide or other intensification agent during this time - bicalutamide is permitted
* Patients may have received palliative radiotherapy for symptomatic bone or visceral metastasis, provided they have recovered from all side effects at the time of registration
* Patients may have received prior surgery. For all major surgeries, at least 14days must have elapsed since completion and patient must have recovered from all major side effects of surgery per investigator's assessment
* Patients may have received or plan to receive concurrent bone targeting agents that do not have an effect on prostate specific antigen (PSA) (e.g. denosumab or bisphosphonate)

Exclusion Criteria:

* Patients must not have received prior and/or must not have any plans for receiving concomitant therapy with ketoconazole, aminoglutethimide, or enzalutamide (MDV3100). Concurrent megestrol for hot flashes is allowed
* Patients must not have received any prior cytotoxic chemotherapy for metastatic prostate cancer

  * Prior cytotoxic chemotherapy with curative intent in the neoadjuvant or adjuvant setting may be allowed at the discretion of the principal investigator. At least 2 years must have elapsed since completion of cytotoxic chemotherapy in the neoadjuvant and/or adjuvant setting
* Patients with known brain metastases are not eligible. Brain imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms suggestive of brain metastasis. But, if brain imaging studies are performed, they must be negative for disease
* Patients must not have New York Heart Association class III or IV heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction, or serious uncontrolled cardiac arrhythmia within 6 months prior to registration
* Patients must not have uncontrolled hypertension (defined as blood pressure > 160 mmHg systolic and > 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart) despite appropriate medical therapy. Note: Patients may be rescreened after adjustments of antihypertensive medications
* Patients must not be known to have human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study
* Patients with a known history of primary and secondary adrenal insufficiency are not eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the study drugs
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy. Previous experimental therapy must have been completed at least 28 days prior to registration
* Patients must not have known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of any of the study drugs, including difficulty swallowing oral medications
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA) nadir < 0.2 | At 12 months
  Will be estimated with 95% Clopper-Pearson interval.

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be determined using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for patients with measurable disease only, and summarized by % of patients achieving complete response, partial response, stable disease, or progressive disease as best response.
PSA responses | Up to 2 years
  Will be described by waterfall plots as recommended by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) as well as identifying the % of patients achieving a 50% and 90% reduction in PSA.
Radiographic progression-free survival (PFS) | Up to 2 years
  Will be evaluated for all patients, using RECIST for soft tissue and including the PCWG3 criteria for bone scan assessment of progression of disease. PFS will be carried out by Kaplan-Meier curve and log-rank test will be used to detect difference between groups.
Patient reported outcomes | Up to 2 years
  Will be collected using Functional Assessment of Cancer Therapy- Prostate and evaluated for changes from baseline, endpoint will be time to deterioration in quality of life.
Androgen receptor (AR) genetic variations | Up to 2 years
  The effect of AR genetic variations on PSA nadir <0.2 at 12 months, ORR, PSA response or PFS. AR CAG and GGC repeats will be analyzed as a continuous variable as well dichotomized as high versus low. PSA nadir results will be compared between CAG/GGC repeat groups.

OTHER OUTCOMES:
Circulating tumor deoxyribonucleic acid (ctDNA) | At baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States